CLINICAL TRIAL: NCT03631004
Title: Pre-operative Olanzapine as Prophylactic Antiemetic in Oncologic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1287/18
Record Dates: First submitted 2018-08-11; First posted 2018-08-15 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Nausea; Postoperative Nausea and Vomiting
Keywords: nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Olanzapine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- olanzapine tablets (Experimental): PATIENT WILL TAKE OLANZAPINE 10 MG, 1 hour BEFORE SURGERY
  Interventions: Drug: Olanzapine
- Starch tablets (Placebo Comparator): PATIENT WILL TAKE PLACEBO 1 hour BEFORE SURGERY
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — olanzapine 10 mg is given before surgery
  Other Names: Treatment

SUMMARY:
Olanzapine has been used as prophylactic antiemetic for chemotherapy induced nausea and vomiting.

The project aims to evaluate the efficacy of olanzapine in combination with ondansetron and dexamethasone in patients at high risk of postoperative nausea and vomiting, with previous history of nausea and vomiting induced by prior chemotherapy, submitted to medium and large surgery.

DETAILED DESCRIPTION:
Double blinded randomized clinical trial. Fifty patients will be selected for each group. Group A will receive 10mg olanzapine in the preoperative and group B will receive placebo in the preoperative period. Both groups will receive intravenous general anesthesia combined with epidural. All patients will receive epidural PCA.

The primary outcome of this study is the incidence of post-operative nausea and vomiting. The power of analysis was based on the following parameters: type error I (α = 0.05), error II (β = 0.8), 95% confidence interval and hypothesis test two-tailed. Thus, 42 patients are indicated per group to obtain reduction of the incidence of nausea and / or vomiting of the population risk from 60% to 30%. The population will be composed of 100 patients because it is assumed that percentage of loss of 10% per group.

The statistical analysis will be performed in program R version 3.5.1. The results obtained will be presented as mean + standard deviation for continuous data or absolute frequency for described data.

For quantitative variables, the Student's t-test will be used for with normal distribution or Mann-Whitney for non-distributed data normal.

For qualitative variables, the chi-square test will be used or Fisher's exact test. Significant difference is defined as p, 0.05.

Data will be collected and managed using REDCap data capture tools

ELIGIBILITY:
Inclusion criteria:

* Patients submitted to medium and large surgeries in the thoracic or abdominal region (mastectomies, breast plastic, hysterectomies, annexectomies, gynecological pelvic surgeries, colectomies, rettosigmoidectomies) under general anesthesia
* Patients aged between 18 and 60 years
* Patients considered to be at high risk for PONV according to the Apfel scale (Apfel 3 or 4)
* Patients with a history of chemotherapy-induced nausea and vomiting.

Exclusion criteria:

* Pregnancy or Lactation
* Current use of typical anti-psychotic medications or atypical
* History of allergy to olanzapine
* Myocardial infarction or unstable angina in the 6 months prior to the day of surgery planning
* History of severe ventricular arrhythmia (eg, VT or VF)
* Heart Failure Class II or greater second NYHA
* Postural hypotension or vasovagal syncope in the 6 months prior to the day of surgery planning
* Narrow angle glaucoma
* Parkinson's disease
* Dementia
* Inability to swallow medicines
* QT interval history greater than 450ms or torsades de pointes
* Patient does not want to participate in the study
* Videolaparoscopy surgery
* Contraindication for neuraxial block

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | 0-24 hours
  nausea and vomiting/ retching (dichotomous variable)

SECONDARY OUTCOMES:
incidence of side effects | 0-6 hours
  side effects
incidence of side effects | 0-24 hours
  side effects
incidence of side effects | 24-48 hours
  side effects
incidence of postoperative nausea and vomiting | 0-6 hours
  nausea and vomiting/ retching (dichotomous variable)
incidence of postoperative nausea and vomiting | 24-48 hours
  nausea and vomiting/ retching (dichotomous variable)
incidence of postoperative nausea | 0-6 hours
  nausea and vomiting/ retching (dichotomous variable)
incidence of postoperative nausea | 0-24 hours
  nausea and vomiting/ retching (dichotomous variable)
incidence of postoperative nausea | 24-48 hours
  nausea and vomiting/ retching (dichotomous variable)
incidence of postoperative vomiting/retching | 0-6 hours
  vomiting/ retching (dichotomous variable)
incidence of postoperative vomiting/retching | 0-24 hours
  vomiting/ retching (dichotomous variable)
incidence of postoperative vomiting/retching | 24-48 hours
  vomiting/ retching (dichotomous variable)
incidence of severe PONV | 0-6 hours
  This scale consists of four questions. Each question generates a different score. For the first question, if the patient vomited or retched three or more times, the final score was 50. Otherwise, the highest score from question 1 or question 2 was multiplied by the scores of question 3 and question 4, yielding the final value. When the score was ≥ 50, the symptom was considered clinically important.
incidence of severe PONV | 0-24 hours
  This scale consists of four questions. Each question generates a different score. For the first question, if the patient vomited or retched three or more times, the final score was 50. Otherwise, the highest score from question 1 or question 2 was multiplied by the scores of question 3 and question 4, yielding the final value. When the score was ≥ 50, the symptom was considered clinically important.
incidence of severe PONV | 24-48 hours
  This scale consists of four questions. Each question generates a different score. For the first question, if the patient vomited or retched three or more times, the final score was 50. Otherwise, the highest score from question 1 or question 2 was multiplied by the scores of question 3 and question 4, yielding the final value. When the score was ≥ 50, the symptom was considered clinically important.
incidence of nausea severity | 0-6 hours
  mild, moderate, or severe
incidence of nausea severity | 0-24 hours
  mild, moderate, or severe
incidence of nausea severity | 24-48 hours
  mild, moderate, or severe

CONTACTS AND LOCATIONS:
Overall Officials: Roger Chammas, Study Director — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Cancer Institute of the State of Sao Paulo - ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No